CLINICAL TRIAL: NCT07077746
Title: A Randomized, Double-Blind, Phase 2, Efficacy and Safety Study of Allogeneic HB-adMSCs vs Placebo for the Treatment of Crohn's Disease
Brief Title: HB-adMSCs for the Treatment of Crohn's Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hope Biosciences Research Foundation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HBCD01
Record Dates: First submitted 2025-07-08; First posted 2025-07-22 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Crohn Disease (CD)
Keywords: Crohn's; Crohn's Disease; Autoimmune; CD; IBD; Inflammatory bowel disease; biologic; stem cell
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: This study is a randomized, double-blind, phase 2, efficacy and safety study of allogeneic HB-adMSCs vs placebo for the treatment of Crohn's Disease. This clinical trial includes a screening period (up to 35 days), a 16-week treatment period and a safety and efficacy follow up period for 52 weeks post first treatment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This clinical trial is a double-blinded study, meaning that the subjects and the researchers both do not know the group assignments. Research staff and subjects may be unblinded once all study data has been collected, all study-related procedures and follow-ups are completed, and all monitoring has been completed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Allogeneic adipose-derived HB-adMSCs (Experimental): Allogeneic HB-adMSCs (Hope Biosciences adipose derived mesenchymal stem cells), Intravenous
  Interventions: Drug: HB-adMSCs - Hope Biosciences Adipose Derived Mesenchymal Stem Cells
- 0.9% sodium chloride (Placebo Comparator): 0.9% sodium chloride, Intravenous
  Interventions: Drug: 0.9% sodium chloride

INTERVENTIONS:
Drug: HB-adMSCs - Hope Biosciences Adipose Derived Mesenchymal Stem Cells — Allogeneic HB-adMSCs (Hope Biosciences adipose derived mesenchymal stem cells). Dose: 200 million cells (+/- 20%) suspended in 20mL 0.9% sodium chloride. Route: Intravenous. Regimen: Weeks 0, 2, 4, 8, 12, and 16. Preparation: HB-adMSCs syringe should be diluted in 250 mL 0.9% sodium chloride (for a total volume of 270 mL).
  Arms: Allogeneic adipose-derived HB-adMSCs
Drug: 0.9% sodium chloride — 0.9% sodium chloride Dose: N/A - 20mL 0.9% sodium chloride. Route: Intravenous. Regimen: Weeks 0, 2, 4, 8, 12, and 16. Preparation: Placebo syringe should be diluted in 250 mL 0.9% sodium chloride (for a total volume of 270 mL).
  Arms: 0.9% sodium chloride

SUMMARY:
Methodology: Randomized, double-blind, efficacy and safety study of allogeneic HB-adMSCs vs placebo for the treatment of Crohn's Disease with a 16-week treatment period and a safety and efficacy follow up period for 52 weeks post first treatment.

Treatment Duration: 16 weeks

General Objectives: To assess the efficacy and safety of multiple intravenous infusions of allogeneic HB-adMSCs by improving signs and symptoms of Crohn's Disease in this subject population.

Number of Subjects: 46 (23 in each treatment arm)

Indication: Crohn's Disease

DETAILED DESCRIPTION:
Primary Objective:

- To investigate the efficacy of intravenous infusions of allogeneic HB-adMSCs vs placebo in patients with Crohn's Disease as determined by improvements in Crohn's Disease Activity Index (CDAI) scores. (Time Frame: Week 0 to Week 52). Minimal clinically important difference (MCID) for CDAI is defined as a decrease of ≥100 points.

Secondary Objectives:

* To assess the safety of intravenous infusions of allogeneic HB-adMSCs vs placebo in patients with Crohn's Disease as determined by the incidence of adverse events or serious adverse events. (Time Frame: Week 0 to Week 52).
* To evaluate the efficacy of intravenous infusions of allogeneic HB-adMSCs vs placebo in patients with Crohn's Disease as determined by improvements in fecal calprotectin (FC) values. (Time Frame: Week 0 to Week 52). Clinically significant changes in fecal calprotectin (FC) values are defined as a ≥50% reduction in fecal calprotectin concentration from baseline, or a decrease to <250 µg/g, whichever is achieved first.

Exploratory Objectives:

* To evaluate the efficacy of intravenous infusions of allogeneic HB-adMSCs vs placebo in patients with Crohn's Disease as determined by improvements in CRP values. (Time Frame: Week 0 to Week 52).
* To evaluate the efficacy of intravenous infusions of allogeneic HB-adMSCs vs placebo in patients with Crohn's Disease as determined by improvements in ESR values. (Time Frame: Week 0 to Week 52).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects who are ≥ 18 years old and ≤ 65 years old.
2. Must be diagnosed with Crohn's Disease at least 6 months prior to the screening visit, as verified by one or more of the following diagnostic criteria present in the participant's medical records:

   1. Clinical presentation of symptoms such as diarrhea, abdominal pain, weight loss, fever, and fatigue
   2. Radiologic Findings within 3 years of screening date: Imaging studies like CT scans or MRI scans of the abdomen and pelvis that indicate bowel wall thickening, strictures, fistulas, and abscesses characteristic of Crohn's disease
   3. Histologic Findings within 3 years of screening date: Microscopic examination of tissue biopsies that indicate transmural inflammation with lymphoid infiltrates
   4. Exclusion of other conditions: Differential diagnoses, such as ulcerative colitis, infectious enterocolitis, and drug-induced colitis, must be excluded through appropriate evaluation
3. Must have CDAI scores at the screening visit of ≥ 150 to ≤ 450, indicating Mild or Moderate Crohn's Disease.
4. Subjects without a current established treatment for Crohn's Disease, or if being treated, subjects who are on a stable dose of Crohn's Disease therapy regimen for ≥3 months prior to screening.
5. Subjects must be willing to maintain their established treatment for Crohn's Disease (or lack thereof) for the duration of the study. Subjects must acknowledge that they may be removed from participation in the study for failure to maintain their established treatment for Crohn's Disease (or lack thereof).
6. Subjects must have an elevated CRP value at the screening visit of ≥1 mg/L and/or an abnormal ESR value at the screening visit of > 15 mm/hr. for male subjects or > 20 mm/hr. for female subjects.
7. Subjects must be able to provide the latest (specifically, within 3 years of screening date) diagnostic imaging records for their Crohn's Disease (including but not limited to endoscopy, colonoscopy, MRI scans, ultrasounds, etc.)
8. Female study subjects of childbearing potential should not be pregnant or plan to become pregnant during study participation and for 6 months after the last investigational product administration. Female study subjects of childbearing potential must confirm usage of one of the following contraceptive measures:

   1. Hormonal contraceptives associated with ovulation inhibition (oral, injectable, implantable, patch, or intravaginal).
   2. Intrauterine device (IUD), or intrauterine hormone-releasing system (IUS).
   3. Barrier contraceptive methods (condoms, diaphragm, etc.). OR Male subjects if their sexual partners can become pregnant should ensure the use one of the following methods of contraception during study participation and for 6 months after the last administration of the investigated product:.

   <!-- -->

   1. Hormonal contraceptives associated with ovulation inhibition (oral, injectable, implantable, patch, or intravaginal).
   2. Intrauterine device (IUD), or intrauterine hormone-releasing system (IUS).
   3. Barrier contraceptive methods (condoms, diaphragm, etc.).
9. Study subjects are able and willing to comply with the requirements of this clinical trial.
10. Voluntarily signed informed consent from study subject or legally authorized representative obtained before any clinical-trial related procedures are performed.

Exclusion Criteria:

1. Study subject has any of the following laboratory results at the screening visit:

   1. WBC: <3000 cells/μL OR >15000 cells/μL (<3 K cells/μL or >15 K cells/μL)
   2. Absolute Neutrophil Count: <1500 cells/μL
   3. Sodium: <120 mEq/L OR >150 mEq/L
   4. Glucose: >150 mg/dL (for fasting subjects)
   5. Potassium: <3.5 mEq/L OR >6 mEq/L
   6. BUN: >25 mg/dL
   7. Creatinine: >2 mg/dL
   8. BUN/Creatinine ratio: >50
2. Study subject has CDAI scores of < 150 or > 450 at the screening visit.
3. Study participant has any vital sign abnormalities at the screening visit as determined by the investigator.
4. Study subject has any of the following cardiovascular issues:

   1. Severe heart failure (e.g., NYHA Class III/IV)
   2. Uncontrolled arrhythmias
   3. Recent myocardial infarction (<6 months from screening visit)
   4. Uncontrolled hypertension
5. Study Subject has any of the following pulmonary diseases:

   1. Severe COPD
   2. Pulmonary fibrosis
   3. History of recent (<6 months from screening visit) pulmonary embolism or DVT
6. Study subject has 1 or more significant uncontrolled concurrent medical conditions (verified by medical records), including the following:

   1. Diabetes Mellitus
   2. Rheumatoid Arthritis
   3. Lupus
   4. Multiple Sclerosis
7. Study subject has any active malignancy, including evidence of cutaneous basal, squamous cell carcinoma or melanoma.
8. Study subject has a history of cancer within 5 years of screening visit (unless curatively treated and without recurrence)
9. Study subject has known alcoholic addiction or dependency or has current substance use or abuse.
10. Receiving any investigational therapy or any approved therapy for investigational use within 1 year prior first dose of the investigational product other than COVID-19 vaccines.
11. Study subject has any other laboratory abnormality or medical condition which, in the opinion of the investigator, poses a safety risk or will prevent the subject from completing the study.
12. Study subject unable to understand and provide signed informed consent.
13. Study subject unlikely to complete the study or adhere to the study procedures.
14. Study subject with known concurrent acute or chronic viral hepatis B or C or human immunodeficiency virus (HIV) infection.
15. Study subject with any systemic infection requiring treatment with antibiotics, antivirals, or antifungals within 30 days prior to first dose of the investigational product.
16. Female subjects who plan to donate eggs or undergo in vitro fertilization treatment during the study within 6 months after the last infusion. OR Male subjects who plan to donate sperm during the study within 6 months after the last infusion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Changes from Baseline in Crohns Disease Activity Index (CDAI) Scores. | Week 0 (Visit 1) to Week 52 (Visit 9)
  Changes from Baseline (Week 0) up to Week 52 in Crohn's Disease Activity Index (CDAI) scores.
  Specifically, clinical response defined as a reduction of at least 100 points in Crohn's Disease Activity Index (CDAI) from baseline. Score ranges from 0 (minimum) - 450 (maximum), the least being asymptomatic and the greatest being most severe.

SECONDARY OUTCOMES:
Incidence of serious adverse events (SAEs). | Week 0 (Visit 1) to Week 52 (Visit 9)
  Incidence of serious adverse events (SAEs).
Incidence of treatment-emergent adverse events (TEAEs). | Week 0 (Visit 1) to Week 20 (Visit 8)
  Incidence of treatment-emergent adverse events (TEAEs). Treatment-emergent adverse events are defined as any adverse events which occur after the first treatment (Week 0) up to the Follow Up Visit (Week 20).
Incidence and risk of AEs of particular interest (serious or non serious), including thromboembolic events, infections, and hypersensitivities | Week 0 (Visit 1) to Week 52 (Visit 9)
  Incidence and risk of AEs of particular interest (serious or non serious), including thromboembolic events, infections, and hypersensitivities.
Changes from Baseline in laboratory values results - Complete Blood Count (x10^3 Cells/uL) | Week 0 (Visit 1) to Week 52 (Visit 9)
  Clinically significant changes from Baseline in laboratory values results - Complete Blood Count (x10^3 Cells/uL)
Changes from Baseline in laboratory values results - Complete Blood Count (% of WBC) | Week 0 (Visit 1) to Week 52 (Visit 9)
  Clinically significant changes from Baseline in laboratory values results - Complete Blood Count (% of WBC)
Changes from Baseline in laboratory values results - Complete Blood Count (pg) | Week 0 (Visit 1) to Week 52 (Visit 9)
  Clinically significant changes from Baseline in laboratory values results - Complete Blood Count (pg)
Changes from Baseline in laboratory values results - Complete Blood Count (g/dL) | Week 0 (Visit 1) to Week 52 (Visit 9)
  Clinically significant changes from Baseline in laboratory values results - Complete Blood Count (g/dL)
Changes from Baseline in laboratory values results - Complete Blood Count (fL) | Week 0 (Visit 1) to Week 52 (Visit 9)
  Clinically significant changes from Baseline in laboratory values results - Complete Blood Count (fL)
Changes from Baseline in laboratory values results - Complete Blood Count (x10^6 Cells/uL) | Week 0 (Visit 1) to Week 52 (Visit 9)
  Clinically significant changes from Baseline in laboratory values results - Complete Blood Count (x10^6 Cells/uL)
Changes from Baseline in laboratory values results - Complete Blood Count (% Difference in Volume and Size of RBC) | Week 0 (Visit 1) to Week 52 (Visit 9)
  Clinically significant changes from Baseline in laboratory values results - Complete Blood Count (% Difference in Volume and Size of RBC)
Changes from Baseline in laboratory values results - Complete Blood Count (% of Total Blood Cell Count) | Week 0 (Visit 1) to Week 52 (Visit 9)
  Clinically significant changes from Baseline in laboratory values results - Complete Blood Count (% of Total Blood Cell Count)
Changes from Baseline in laboratory values results - Comprehensive Metabolic Panel (g/dL) | Week 0 (Visit 1) to Week 52 (Visit 9)
  Clinically significant changes from Baseline in laboratory values results - Comprehensive Metabolic Panel (g/dL)
Changes from Baseline in laboratory values results - Comprehensive Metabolic Panel (Ratio of Albumin to Calc. Globulin) | Week 0 (Visit 1) to Week 52 (Visit 9)
  Clinically significant changes from Baseline in laboratory values results - Comprehensive Metabolic Panel (Ratio of Albumin to Calc. Globulin)
Changes from Baseline in laboratory values results - Comprehensive Metabolic Panel (U/L) | Week 0 (Visit 1) to Week 52 (Visit 9)
  Clinically significant changes from Baseline in laboratory values results - Comprehensive Metabolic Panel (U/L)
Changes from Baseline in laboratory values results - Comprehensive Metabolic Panel (mg/dL) | Week 0 (Visit 1) to Week 52 (Visit 9)
  Clinically significant changes from Baseline in laboratory values results - Comprehensive Metabolic Panel (mg/dL)
Changes from Baseline in laboratory values results - Comprehensive Metabolic Panel (mEq/L) | Week 0 (Visit 1) to Week 52 (Visit 9)
  Clinically significant changes from Baseline in laboratory values results - Comprehensive Metabolic Panel (mEq/L)
Changes from Baseline in laboratory values results - Comprehensive Metabolic Panel (mL/Min/1.73m^2) | Week 0 (Visit 1) to Week 52 (Visit 9)
  Clinically significant changes from Baseline in laboratory values results - Comprehensive Metabolic Panel (mL/Min/1.73m^2)
Changes from Baseline in laboratory values results - Comprehensive Metabolic Panel (Ratio of Calc BUN/Creatinine) | Week 0 (Visit 1) to Week 52 (Visit 9)
  Clinically significant changes from Baseline in laboratory values results - Comprehensive Metabolic Panel (Ratio of Calc BUN/Creatinine)
Changes from Baseline in laboratory values results - Coagulation Panel (Seconds) | Week 0 (Visit 1) to Week 52 (Visit 9)
  Clinically significant changes from Baseline in laboratory values results - Coagulation Panel (Seconds)
Changes from Baseline in laboratory values results - Coagulation Panel (Ratio of Prothrombin Time/Mean Prothrombin Time) | Week 0 (Visit 1) to Week 52 (Visit 9)
  Clinically significant changes from Baseline in laboratory values results - Coagulation Panel (Ratio of Prothrombin Time/Mean Prothrombin Time)
Changes from Baseline in Vital Signs - Respiratory Rate (Breaths per minute) | Week 0 (Visit 1) to Week 52 (Visit 9)
  Clinically significant changes from baseline in Respiratory Rate (Breaths per minute)
Changes from Baseline in Vital Signs - Heart Rate (Breaths per minute) | Week 0 (Visit 1) to Week 52 (Visit 9)
  Clinically significant changes from baseline in Heart Rate (Breaths per minute)
Changes from Baseline in Vital Signs - Body Temperature (Celsius) | Week 0 (Visit 1) to Week 52 (Visit 9)
  Clinically significant changes from baseline in Body Temperature (Celsius)
Changes from Baseline in Vital Signs - Systolic Blood Pressure (mmHg) | Week 0 (Visit 1) to Week 52 (Visit 9)
  Clinically significant changes from baseline in Systolic Blood Pressure (mmHg)
Changes from Baseline in Vital Signs - Diastolic Blood Pressure (mmHg | Week 0 (Visit 1) to Week 52 (Visit 9)
  Clinically significant changes from baseline in Diastolic Blood Pressure (mmHg)
Changes from Baseline in Vital Signs - SPO2 (%) | Week 0 (Visit 1) to Week 52 (Visit 9)
  Clinically significant changes from baseline in SPO2 (%)
Clinically significant changes in Weight results (in kg) | Week 0 (Visit 1) to Week 52 (Visit 9)
  Clinically significant changes in weight (kg)
Number of participants with abnormal physical examination results - Abdomen | Week 0 (Visit 1) to Week 52 (Visit 9)
  Number of participants with abnormal physical examination results - Abdomen
Number of participants with abnormal physical examination results - Cardiovascular | Week 0 (Visit 1) to Week 52 (Visit 9)
  Number of participants with abnormal physical examination results - Cardiovascular
Number of participants with abnormal physical examination results - Head, Eyes, Ears, Nose, and Throat | Week 0 (Visit 1) to Week 52 (Visit 9)
  Number of participants with abnormal physical examination results - Head, Eyes, Ears, Nose, and Throat
Number of participants with abnormal physical examination results - Lymph Node | Week 0 (Visit 1) to Week 52 (Visit 9)
  Number of participants with abnormal physical examination results - Lymph Node
Number of participants with abnormal physical examination results - Musculoskeletal | Week 0 (Visit 1) to Week 52 (Visit 9)
  Number of participants with abnormal physical examination results - Musculoskeletal
Number of participants with abnormal physical examination results - Neurological | Week 0 (Visit 1) to Week 52 (Visit 9)
  Number of participants with abnormal physical examination results - Neurological
Number of participants with abnormal physical examination results - Respiratory | Week 0 (Visit 1) to Week 52 (Visit 9)
  Number of participants with abnormal physical examination results - Respiratory
Number of participants with abnormal physical examination results - Skin | Week 0 (Visit 1) to Week 52 (Visit 9)
  Number of participants with abnormal physical examination results - Skin
Change from Baseline in Fecal Calprotectin (FC) values. | Week 0 (Visit 1) to Week 52 (Visit 9)
  Clinically significant changes in Fecal Calprotectin (FC) values, defined as a ≥50% reduction in fecal calprotectin concentration from baseline, or a decrease to <250 µg/g, whichever is achieved first.

OTHER OUTCOMES:
Change from Baseline in C-Reactive Protein values. | Week 0 (Visit 1) to Week 52 (Visit 9)
  Clinically significant changes in C-Reactive Protein values.
Change from Baseline in erythrocyte sedimentation rate values. | Week 0 (Visit 1) to Week 52 (Visit 9)
  Clinically significant changes in erythrocyte sedimentation rate values.

CONTACTS AND LOCATIONS:
Overall Officials: Thanh Cheng, MD, Principal Investigator — Hope Biosciences Research Foundation
Locations (1):
- Hope Biosciences Research Foundation, Sugar Land, Texas, United States